CLINICAL TRIAL: NCT05084768
Title: Integration of Donor-derived Cell-free DNA With HLA-DR+TNFR2+ Regulatory T Cell in the Prediction of Acute Rejection and Graft Function After Kidney Transplantation
Brief Title: Dd-cfDNA and Treg in Prediction of Kidney Transplant Acute Rejection
Status: Recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5210340
Record Dates: First submitted 2021-09-18; First posted 2021-10-20 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Acute Rejection of Renal Transplant; Graft Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rejection of kidney transplant: Diagnostic test: measurement of regulatory T cell and donor-derived cell-free DNA
  Interventions: Diagnostic Test: Donor-derived cell-free DNA
- No rejection of kidney transplant: Diagnostic test: measurement of regulatory T cell and donor-derived cell-free DNA
  Interventions: Diagnostic Test: Donor-derived cell-free DNA

INTERVENTIONS:
Diagnostic Test: Donor-derived cell-free DNA — As mentioned previously
  Other Names: Regulatory T cell

SUMMARY:
Acute rejection after kidney transplantation should ideally be diagnosed prior to immunologic injury in a non-invasive fashion in order to improve long-term graft function. Donor-derived cell-free DNA (ddcfDNA) is a promising method to do so as it is elevated prior to acute rejection and has good predictive performance especially for antibody-mediated and high severity T-cell mediated rejection. Its ability to predict low severity T-cell mediated rejection and future graft function remains equivocal. Regulatory T cells (Tregs) are essential in transplant tolerance by suppressing effector immune responses. Circulating post-transplant highly suppressive HLA-DR+ Tregs were reduced in recipients who developed acute rejection. Preliminary results in a cohort including predominantly low severity T-cell mediated rejection also showed that pre-transplant circulating highly suppressive TNFR2+ Tregs were reduced in and could predict acute rejection. Integrating dd-cfDNA with HLA-DR+TNFR2+ Treg could improve the predictive performance for acute rejection especially of low severity and potentially predict graft function. Plasma dd-cfDNA and HLA-DR+TNFR2+ Tregs will be measured in 150 kidney transplant recipients at scheduled intervals during the first 6 months post-transplant. Predictive accuracy of a model integrating ddcfDNA and HLA-DR+TNFR2+ Treg for acute rejection will be tested using ROC curve analysis and multivariate logistic regression. Predictive accuracy for 1-year graft function will be tested using multivariate linear regression. High predictive performance for acute rejection and graft function using a model integrating dd-cfDNA and HLA-DR+TNFR2+ Treg would help identify kidney transplant recipients at immunologic risk early on and allow personalization of immunosuppression accordingly.

DETAILED DESCRIPTION:
Background

Despite advances in immunosuppression, 10-year graft survival after kidney transplantation has remained stagnant at around 50%. Timely diagnosis of acute rejection in kidney transplant recipients is essential for improving long-term graft survival. Clinical suspicion for acute rejection currently relies on monitoring elevation in serum creatinine and diagnostic confirmation with a kidney allograft biopsy. Serum creatinine elevation, however, is non-specific for acute rejection and is detected after significant immunological damage to the allograft already happens. Confirmation with a biopsy is invasive, associated with a 1% major complication rate, and subjected to inadequate sampling as well as expert reader variance. Novel ways to monitor and diagnose acute rejection prior to immunological injury in a non-invasive fashion are needed in an effort to improve long-term graft survival after kidney transplantation. Cell-free DNA is normally released into the bloodstream when cells undergo apoptosis or necrosis. In the context of kidney transplantation and the presence of an allograft, donor-derived cell-free DNA (dd-cfDNA) is continuously shed into the bloodstream of the recipient as a result of allograft cell turnover and represents a small fraction of total cell-free DNA (donor- plus recipient-derived). Dd-cfDNA fraction is initially high from ischemia-reperfusion injury and usually decreases to a baseline level 10 to 14 days after kidney transplantation. Subsequently, episodes of allograft injury such as acute rejection leads to an increase in dd-cfDNA fraction into the recipient's bloodstream. Using single-nucleotide polymorphisms-based multiplexed polymerase chain reaction technology and advanced bioinformatics, plasma dd-cfDNA fraction can now be measured in a kidney transplant recipient without the need for prior genotyping of the donor or the recipient. Recent studies have demonstrated that plasma dd-cfDNA is a promising novel method to detect acute rejection prior to immunological injury in a non-invasive fashion as it is elevated in advance and at the time of biopsy-proven acute rejection. A cutoff dd-cfDNA fraction greater or equal to 1% was able to predict acute rejection with moderate to good performance in those studies with area under the curves (AUCs) varying from 0.59 - 0.97 on receiver operating characteristic (ROC) curve analyses. When examining acute rejection by mechanism, dd-cfDNA fraction appears to have better predictive performance for antibody-mediated rejection (ABMR), while its utility to predict T cell-mediated rejection (TCMR) remains equivocal especially when of lower severity (less than Banff 1B). Nevertheless, in lower severity TCMR (Banff 1A or subclinical), a dd-cfDNA fraction greater or equal to 0.5% was shown to potentially identify kidney transplant recipients at risk for a steeper estimated glomerular filtration rate (eGFR) decline, developing de-novo donor specific antibody, and future rejection episodes. Despite being approved for clinical use by Medicare, several limitations remain with dd-cfDNA in the prediction of acute rejection. First, elevation in dd-cfDNA is not rejection-specific as other medical complications such as urinary tract infections, systemic infections, and BK virus nephropathy can also increase dd-cfDNA. Secondly, predictive performance of dd-cfDNA for TCMR, especially of lower severity, remains equivocal. Finally, it is unclear whether early dd-cfDNA fraction after kidney transplantation can predict future immunologic graft injuries and function. Novel ways to make dd-cfDNA more specific for acute rejection, improve its predictive performance for TCMR, and correlate it with future graft function would further improve its clinical utility. Regulatory T cells (Tregs) are essential in the induction and maintenance of tolerance in various kidney transplant animal models by suppressing effector immune responses. Tregs constitute 5 - 10% of CD4+ T cells and are traditionally identified as a homogeneous population with high expression of CD25, low expression of CD127, and expression of the master transcription factor FoxP3. Recent data, however, indicate that Tregs are more heterogeneous and that expression of additional molecules than the traditional CD25, CD127, and FoxP3 influence their suppressive functional activity. In human kidney transplantation, posttransplant circulating CD4+CD25hiCD127lo/- Tregs were similar between recipients who suffered from acute rejection and those that did not. However, high expression of HLA-DR on post-transplant circulating Tregs, which identified a population with maximally suppressive functional activity, was lower in recipients who suffered from acute rejection. Another molecule identifying a Treg population with maximally suppressive functional activity is TNFR2. TNFR2 mediates the biological function of the pro-inflammatory cytokine TNF-a, which is involved in the recruitment and activation of effector T cells during allograft rejection. Interestingly, TNFR2 was shown to be preferentially expressed on Tregs as opposed to effector T cells. In both murine and human studies, TNF-α signaling via TNFR2+ Tregs increased their survival, proliferation, and suppressive functional activity.

Preliminary results The investigators previously studied TNFR2+ Tregs in the specific context of kidney transplantation. The investigators confirmed in a cohort of kidney transplant candidates that expression of TNFR2 on Tregs correlated with suppressive function measured via a traditional co-culture assay of Tregs with stimulated effector T cells (r=0.63, p<0.01). In a cohort of 76 deceased donor kidney transplant recipients, the investigators published on the role of pre-transplant circulating recipient TNFR2+ Tregs in the prediction of delayed and slow graft function after kidney transplantation. Since delayed and slow graft function are known risk factors for the development of acute rejection after kidney transplantation, the investigators then examined the role of pre-transplant circulating recipient TNFR2+ Tregs in the prediction of acute rejection in the same cohort of recipients in which 75 had available acute rejection data with promising results especially with low severity TCMR.

Hypotheses

Since previous studies and the investigators' preliminary results in a cohort predominantly including low severity TCMR suggest a role for HLA-DR+TNFR2+ Tregs in the prediction of acute rejection, the investigators hypothesize that integrating it with dd-cfDNA fraction could improve specificity and predictive performance for acute rejection, especially TCMR. The investigators also hypothesize that measurement of early dd-cfDNA fraction and pretransplant HLA-DR+TNFR2+ Tregs could predict future outcomes after kidney transplantation including acute rejection and graft function measured by eGFR.

Objectives

1. Test whether integrating dd-cfDNA fraction with HLA-DR+TNFR2+ Tregs in advance or at the time of allograft injury can improve the predictive performance for acute rejection after kidney transplantation.
2. Test whether integrating dd-cfDNA fraction at 2 weeks post-transplant with pre-transplant HLADR+TNFR2+ Tregs can predict future acute rejection episodes and 1-year graft function.

The investigators will recruit 150 adult kidney transplant recipients with insurance coverage for dd-cfDNA fraction measurement.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney transplant candidates/recipients

Exclusion Criteria:

* Age less than 18
* Multi-organ transplants
* Kidney transplant candidates/recipients with HIV
* Kidney transplant candidates/recipients with HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult kidney transplant candidates/recipients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with biopsy-proven acute rejection graded with the Banff score | 1 year
  TCMR 1A, TCMR 1B, TCMR 2A, TCMR 2B, TCMR 3B, ABMR

SECONDARY OUTCOMES:
Number of participants with graft failure based on return to chronic dialysis or death | 1 year
  Return to chronic dialysis, Death

CONTACTS AND LOCATIONS:
Overall Officials: Minh-Tri Nguyen, MD PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No